CLINICAL TRIAL: NCT05959915
Title: ECG Monitoring Short vs Middle Term After Atrial Fibrillation Ablation
Acronym: CLARITY
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Josep Lluis Mont Girbau, Head of AF Unit, Hospital Clinic of Barcelona
Other Study IDs: CLARITY
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Device: device e-patch Implantation — The ePatch device (Phillips) was used. This device is attached to the sternum, using a specific dressing adapted for the device itself. Manufacturer's recommendations for skin preparation and placement will be followed.
  The device will remain in place for 4-5 days, at which time the patient will be readmitted for data extraction and reading.
  The team of research nurses will analyze the data through the ePatch platform and later, the electrophysiologists will review the results and make a diagnosis.

SUMMARY:
To compare the number of patients with AF recurrence detected in a 24-h Holter monitoring with a 5-day record.

ELIGIBILITY:
Inclusion Criteria:

* Have undergone an AF ablation procedure at the Hospital Clínic and have a 12-month follow-up planned.
* Having been previously assessed by the AF nurse.
* Having signed the informed consent.

Exclusion Criteria:

* Extreme skin fragility at chest level
* Allergy to latex or adhesive tape
* No electrophysiology follow-up at the Clínic hospital.
* Patients who are already included in other studies that may interfere with the expected results of this one.
* Patients with cognitive impairment or disorientation.

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are evaluated 3 months after having AF ablation surgery.
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
AF recurrence | up to 5 days
  Number of patients with AF recurrence detected in a cardio loop monitoring.

SECONDARY OUTCOMES:
Adverse effects | up to 5 days
  skin injuries, losses, allergies, etc.
Burden of AF | up to 5 days
  Burden of AF in the two groups (Day/Hours/minuts)
Number of patients with recurrent AF / atrial flutter / atrial tachycardia | up to 5 days
  Number of patients with recurrent AF / atrial flutter / atrial tachycardia in two groups
Total time of noise | up to 5 days
  Total time of noise in each group
Total time analized | up to 5 days
  Total time analized in each group
premature losses | up to 5 days
  loss of connection of the device before 5 days
time to analyze | min:hours
  time it takes to analyze and interpret the logs obtained, in minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrade JG, Macle L, Nattel S, Verma A, Cairns J. Contemporary Atrial Fibrillation Management: A Comparison of the Current AHA/ACC/HRS, CCS, and ESC Guidelines. Can J Cardiol. 2017 Aug;33(8):965-976. doi: 10.1016/j.cjca.2017.06.002. Epub 2017 Jun 9. PMID 28754397
- [Background] Forleo GB, Casella M, Dello Russo A, Moltrasio M, Fassini G, Tesauro M, Tondo C. Monitoring Atrial Fibrillation After Catheter Ablation. J Atr Fibrillation. 2014 Apr 30;6(6):1040. doi: 10.4022/jafib.1040. eCollection 2014 Apr-May. PMID 27957062
- [Background] Forkmann M, Schwab C, Edler D, Vevecka A, Butz S, Haller B, Brachmann J, Busch S. Characteristics of early recurrences detected by continuous cardiac monitoring influencing the long-term outcome after atrial fibrillation ablation. J Cardiovasc Electrophysiol. 2019 Oct;30(10):1886-1893. doi: 10.1111/jce.14109. Epub 2019 Aug 26. PMID 31397518
- [Background] Aljuaid M, Marashly Q, AlDanaf J, Tawhari I, Barakat M, Barakat R, Zobell B, Cho W, Chelu MG, Marrouche NF. Smartphone ECG Monitoring System Helps Lower Emergency Room and Clinic Visits in Post-Atrial Fibrillation Ablation Patients. Clin Med Insights Cardiol. 2020 Jan 20;14:1179546820901508. doi: 10.1177/1179546820901508. eCollection 2020. PMID 32009826
- [Background] Kimura T, Aizawa Y, Kurata N, Nakajima K, Kashimura S, Kunitomi A, Nishiyama T, Katsumata Y, Nishiyama N, Fukumoto K, Tanimoto Y, Fukuda K, Takatsuki S. Assessment of atrial fibrillation ablation outcomes with clinic ECG, monthly 24-h Holter ECG, and twice-daily telemonitoring ECG. Heart Vessels. 2017 Mar;32(3):317-325. doi: 10.1007/s00380-016-0866-2. Epub 2016 Jul 6. PMID 27385021
- [Background] Sikorska A, Baran J, Piotrowski R, Krynski T, Szymot J, Soszynska M, Kulakowski P. Daily ECG transmission versus serial 6-day Holter ECG for the assessment of efficacy of ablation for atrial fibrillation - the AGNES-ECG study. J Interv Card Electrophysiol. 2022 Nov;65(2):373-380. doi: 10.1007/s10840-022-01166-4. Epub 2022 Mar 3. PMID 35244820
- [Background] Hermans ANL, Gawalko M, Pluymaekers NAHA, Dinh T, Weijs B, van Mourik MJW, Vorstermans B, den Uijl DW, Opsteyn L, Snippe H, Vernooy K, Crijns HJGM, Linz D, Luermans JGLM. Long-term intermittent versus short continuous heart rhythm monitoring for the detection of atrial fibrillation recurrences after catheter ablation. Int J Cardiol. 2021 Apr 15;329:105-112. doi: 10.1016/j.ijcard.2020.12.077. Epub 2021 Jan 4. PMID 33412184
- [Background] Hillmann HAK, Soltani S, Mueller-Leisse J, Hohmann S, Duncker D. Cardiac Rhythm Monitoring Using Wearables for Clinical Guidance before and after Catheter Ablation. J Clin Med. 2022 Apr 26;11(9):2428. doi: 10.3390/jcm11092428. PMID 35566556
- [Result] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505